CLINICAL TRIAL: NCT04146922
Title: Switch to Oral Antibiotics in Gram-negative Bacteremia (SOAB); a Randomized, Open-label, Clinical Trial.
Brief Title: Switch to Oral Antibiotics in Gram-negative Bacteremia
Acronym: SOAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRC-01-19-254
Record Dates: First submitted 2019-10-20; First posted 2019-10-31 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2022-03

CONDITIONS: Escherichia Coli Bacteremia; Klebsiella Bacteraemia; Enterobacter Bacteraemia; Serratia Bacteraemia; Citrobacter Bacteraemia; Proteus Bacteraemia
Keywords: Enterobacteriaceae, bacteremia, step down oral therapy
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Intervention Model Description: Computer generated block randomization into permuted blocks of 4, 6 and 8
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IV Group (Active Comparator): Eligible patients randomized to complete their antimicrobial therapy course through intravenous (IV) administration.
  Interventions: Other: IV antimicrobial therapy
- Oral Group (Experimental): Eligible patients randomized to step down to oral antimicrobial therapy for the remainder of their treatment course.
  Interventions: Other: Step down to oral antimicrobial therapy

INTERVENTIONS:
Other: Step down to oral antimicrobial therapy — Step down from intravenous to oral antimicrobial therapy to complete the intended course of treatment.
  Arms: Oral Group
Other: IV antimicrobial therapy — No step down from intravenous to oral antimicrobial therapy to complete the intended course of treatment.
  Arms: IV Group

SUMMARY:
Eligible subjects will be those age 18 years or more with mono-microbial blood stream infection caused by E. coli, Klebsiella species, Enterobacter species, Serratia species, Citrobacter species, or Proteus species, who have achieved adequate source control, are afebrile and hemodynamically stable for 48 hours or more and have received microbiologically active intravenous therapy for 3-5 days. The bloodstream isolate must be susceptible to amoxicillin, amoxicillin-clavulanate, fluoroquinolones, oral cephalosporins and/or trimethoprim-sulfamethoxazole and the subject must be able to take oral medication directly or through a feeding tube. Exclusions criteria include allergy to all in-vitro active antimicrobials which are available in oral formulations, pregnancy, infective endocarditis, central nervous system infection, terminal illness with expected survival less than 14 days, absolute neutrophil count less than 1,000/ml and hematopoietic or solid organ transplantation within the preceding 90 days. Randomization will be stratified by urinary versus non-urinary source of bacteremia. The primary outcome is treatment failure at 90-days with 10% margin for non-inferiority in the 95% confidence interval around the difference in outcome between the two study groups.

DETAILED DESCRIPTION:
Oral antimicrobial therapy mitigates vascular line associated complications such as infection, thrombosis and pain, facilitating early mobilization and discharge and reducing healthcare costs. Efficacy and safety of step-down to oral antimicrobial therapy in patients with Enterobacteriaceae bacteremia has never been confirmed in a randomized clinical trial. The aim of this clinical trial is to evaluate the safety and efficacy of oral step down strategy in patients with Gram-negative blood stream infections.

Eligible subjects will be those age 18 years or more with mono-microbial blood stream infection caused by E. coli, Klebsiella species, Enterobacter species, Serratia species, Citrobacter species, or Proteus species, who have achieved adequate source control, are afebrile and hemodynamically stable for 48 hours or more and have received microbiologically active intravenous therapy for 3-5 days. The bloodstream isolate must be susceptible to amoxicillin, amoxicillin-clavulanate, fluoroquinolones, oral cephalosporins and/or trimethoprim-sulfamethoxazole and the subject must be able to take oral medication directly or through a feeding tube. Exclusions criteria include allergy to all in-vitro active antimicrobials which are available in oral formulations, pregnancy, infective endocarditis, central nervous system infection, terminal illness with expected survival less than 14 days, absolute neutrophil count less than 1.0x109/L and hematopoietic or solid organ transplantation within the preceding 90 days.

The primary endpoint is treatment failure at 90-days, defined as a composite of the death from any cause, need for additional antimicrobial therapy with one or more microbiologically active agents before complete resolution of signs and symptoms of infection, microbiological relapse (same species from any clinical site) and infection-related re-admission.

Eligible subjects will be randomized using permuted blocks of variable sizes to full intravenous antimicrobial therapy course (IV Group) or intravenous followed by step-down to oral therapy (PO Group). Randomization will be stratified by urinary versus non-urinary source of bacteremia. The primary analysis will include all patients who were randomized and received at least one dose of the assigned treatment. The difference in primary outcome rate between the intervention and control groups will be presented alongside a 95% confidence interval (CI), adjusted by source of bacteremia. If the upper limit of the 95% CI for the difference in overall response is below 10%, non-inferiority will be concluded.

A Data and Safety Monitoring Board will oversee the trial. An interim analysis will be performed after the first 50% of the target sample have completed the 90-day study period. The Data and Safety Monitoring Board can make a binding recommendation to terminate the study if the results of the interim analysis indicate very high likelihood for positive effect or futility.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Mono-microbial blood stream infection.
* Isolation of E. coli, Klebsiella species, Enterobacter species, Serratia species, Citrobacter species, or Proteus species from ≥1 blood culture(s).
* Adequate source control within ≤5 days of staring in-vitro active intravenous antimicrobial therapy.
* Afebrile (Tmax <38 degrees Celsius) for ≥48 hours.
* Hemodynamically stable for ≥48 hours (SBP ≥100 mmHg, no vasopressors).
* Microbiologically active intravenous therapy for 3-5 days.
* Bloodstreams isolate in-vitro susceptibility to amoxicillin, amoxicillin-clavulanate, fluoroquinolones, oral cephalosporins and/or trimethoprim-sulfamethoxazole.
* Ability to take oral medication directly or through a feeding tube.

Exclusion Criteria:

* Allergy to all in-vitro active antibiotics which are available in oral formulations.
* Pregnancy.
* Infective endocarditis.
* Central nervous system infection.
* Terminal illness with expected survival <14 days.
* Neutropenia (absolute neutrophil count <1.0x10^9/L).
* Hematopoietic or solid organ transplantation within the preceding 90 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2019-10-13 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Treatment failure. | 90 days
  Defined as death, need for additional active antibiotic therapy before resolution of all signs and symptoms of infection, microbiological relapse or infection-related re-admission within 90 days of commencement of active intravenous antimicrobial therapy.

SECONDARY OUTCOMES:
Death from any cause. | 90 days
  Death from any cause during follow up period.
Need for additional antimicrobial therapy with one or more microbiologically active agents before complete resolution of signs and symptoms of infection. | Up to 90 days
  Need for additional active antimicrobial therapy before resolution of signs and symptoms of infection; defined as recovery from infection-related symptoms present at baseline (e.g.; urinary symptoms, abdominal pain, jaundice ..etc), no recurrence of fever (Tmax ≥38.0oC).
Microbiological relapse. 4) | 90 days
  Active infection in any site caused by the same species in the index blood culture.
Infection-related re-admission. | 90 days
  Re-admission to hospital because of any active infection.
Hospital length of stay from date of first positive blood culture. | Up to 90 days
  Hospital length of stay from date of first positive blood culture.

CONTACTS AND LOCATIONS:
Overall Officials: Ali S Omrani, FRCP FRCPath, Study Director — Hamad Medical Corporation
Locations (7):
- Bahrain Defense Forces Hospital, Manama, Bahrain
- Farwaniya Hospital, Kuwait City, Kuwait
- Hamad Medical Corporation, Doha, Qatar
- Turkey (Türkiye) (4):
  - Istanbul Medipol University, Istanbul
  - Istanbul University Carrahpasa Medical School, Istanbul
  - Marmara University School of Medicine, Istanbul
  - Ordu University School of Medicine, Ordu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Omrani AS, Abujarir SH, Ben Abid F, Shaar SH, Yilmaz M, Shaukat A, Alsamawi MS, Elgara MS, Alghazzawi MI, Shunnar KM, Zaqout A, Aldeeb YM, Alfouzan W, Almaslamani MA; SOAB Study Group. Switch to oral antibiotics in Gram-negative bacteraemia: a randomized, open-label, clinical trial. Clin Microbiol Infect. 2024 Apr;30(4):492-498. doi: 10.1016/j.cmi.2023.10.014. Epub 2023 Oct 18. PMID 37858867